CLINICAL TRIAL: NCT07261839
Title: Effect of Visualized Meditation on Anxiety, Pain, and Comfort in Patients Undergoing Endoscopy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Tuğba Albayram, Research Assistant Dr, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/408
Record Dates: First submitted 2025-11-15; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Endoscopy; Pain; Comfort; Randomized Controlled Trial
Keywords: Endoscopy, pain, comfort, visualized meditation; Endoscopy; Pain; Comfort; Visualized meditation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visualized meditation group (Active Comparator): Visualized meditation for patients who have had an endoscopy
  Interventions: Other: Visualized meditation
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: Visualized meditation — In the study, the experimental group will listen to visualized meditation sessions daily, morning and evening, for three days before the endoscopy. On the morning of the endoscopy, patients will be administered a personal information form, STAI1-2, pain scale, and comfort scale. After the procedure, the patients will be taken to the recovery area and will be administered the STAI1-2, pain scale, and comfort scale again.
  Arms: Visualized meditation group

SUMMARY:
Endoscopy is one of the most frequently performed procedures for the early diagnosis and treatment of many diseases and plays a crucial role in the diagnosis and treatment of upper gastrointestinal disorders. Sometimes, endoscopy may be the only option for detecting certain diseases of the stomach and larynx. However, for many patients, endoscopy is considered an invasive, highly painful, and extremely uncomfortable procedure. Furthermore, anxiety and fear felt before the procedure can cause physical and emotional discomfort, disrupt patient comfort, and cause pain.

DETAILED DESCRIPTION:
Endoscopy is one of the most frequently performed procedures for the early diagnosis and treatment of various gastrointestinal disorders and plays a critical role, particularly in the evaluation of upper gastrointestinal system pathologies. In certain clinical situations, endoscopy may be the only reliable method for identifying diseases occurring in the stomach, esophagus, and larynx. Despite its diagnostic and therapeutic value, endoscopy is commonly perceived by patients as an invasive, uncomfortable, and often painful procedure. In addition, the anxiety and fear experienced before the procedure can lead to both physical and emotional distress, negatively affecting overall patient comfort and potentially intensifying the perception of pain.

Moderate to severe anxiety during endoscopy has been shown to increase the likelihood of procedural difficulties, prolong the duration of the examination, reduce patient satisfaction, and elevate the risk of complications. These adverse effects highlight the importance of implementing non-pharmacological strategies aimed at reducing anxiety and improving patient comfort. One such approach-guided visualization or visualized meditation-has gained attention as a simple, cost-effective, and patient-friendly method that promotes relaxation, reduces emotional tension, and supports pain management.

Considering the potential of guided visualization to enhance tolerance to the procedure and improve patient experiences, researchers were motivated to explore its effectiveness in this specific population. Therefore, this study was designed to determine the effect of visualized meditation applied to patients undergoing endoscopy on their levels of anxiety, pain, and comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18, with no hearing impairment,
* Students undergoing endoscopy for the first time,
* Not diagnosed with a psychiatric disorder and therefore not on medication,
* Willing to participate in the study

Exclusion Criteria:

* Patients who refused to participate in the study, underwent endoscopy for biopsy, or received deep sedation.
* Patients who volunteered to participate and then wished to withdraw from the study at any stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS Pain and Comfort Scale | From enrollment to the end of treatment at 4 months
  This scale was developed by Price and colleagues (1983). It is used to measure subjective pain and comfort levels. The scale is represented by a 10-cm line representing the lowest and highest pain scores (0: no pain/discomfort, 10: most intolerable pain/discomfort).
The State Trait Anxiety Inventory (STAI) | "From enrollment to the end of treatment at 4 months
  The State Trait Anxiety Inventory (STAI), developed by Spielberger et al. in 1964, will be used to measure anxiety in this study. The scale has two dimensions: the STAI-S, which measures state anxiety, and the STAI-T, which measures trait anxiety. The STAI-S and STAI-T each consist of 20 items. Items 1-40 on the scale measure anxiety in four ways. The lowest score for both dimensions of the scale is 20, and the highest score is 80. As the score increases, the level of anxiety also increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not plan to share your IPD with other researchers.